CLINICAL TRIAL: NCT05752838
Title: Are Primary Outcomes Really Primary? A Questionnaire Survey Study for Exploring Outcomes for Patients With Disc Herniation Reflecting Real Patient Symptoms and Needs
Brief Title: A Questionnaire Survey Study for Exploring Outcomes for Patients With Disc Herniation
Status: Completed | Type: Observational
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: JS-CT-2022-14
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Lumbar Disc Herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diagnosed with LDH and had LDH-related radiating leg pain
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a survey study, and there were no intervention

SUMMARY:
Background: The selection of primary outcomes that reflect the real symptoms and conditions of patients is instrumental in clinical studies on the effectiveness of specific treatment modalities. This study aimed to explore the appropriate outcomes that reflect the real-world needs and concerns of patients with lumbar disc herniation (LDH) and provide a basis for designing related clinical trials.

Methods and Findings: This cross-sectional nationwide web-based survey study was conducted in South Korea in November 2022. Patients who were diagnosed with LDH and had LDH-related radiating leg pain were enrolled. The questionnaire consisted of 5 parts: basic characteristics, disease onset, symptom and severity, priority symptoms for improvement, and important factors in treatment. Overall, 500 patients (100 patients from the each age group) were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed of LDH
* age 19-69 years
* presence of LDH-related symptoms such as pain, numbness, weakness, or tingling in the legs
* agree to informed consent form

Exclusion Criteria:

* severe mental illness and intellectual disabilities that prevented independence in answering the questionnaire

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All 19-69 patients who were diagnosed with LDH and had LDH-related radiating leg in Korea
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
survey basic characteristics | 1 day
disease onset survey | 1 day
symptom and its severity survey | 1 day
priority symptoms for improvement survey | 1 day
important factors in treatment survey | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Medical Foundation, Seoul, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No